CLINICAL TRIAL: NCT02330471
Title: Forced Versus Spray Coagulation in Women Undergoing LLETZ-conization for Cervical Dysplasia: a Randomized Trial
Acronym: CONE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Clemens Tempfer, MD, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONE-1
Record Dates: First submitted 2014-12-27; First posted 2015-01-05 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Uterine Cervical Dysplasia
Keywords: conization; LLETZ; cervical dysplasia; cervical intraepithelial neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spray (Experimental): cervical coagulation using a superficial electrical coagulation mode, ie spray coagulation
  Interventions: Procedure: Spray
- Forced (Active Comparator): cervical coagulation using a deep tissue electrical coagulation mode, ie forced coagulation
  Interventions: Procedure: Forced

INTERVENTIONS:
Procedure: Spray — surgical method to achieve intraoperative hemostasis by a superficial electrocoagulation of 80 Watt voltage
  Arms: Spray
Procedure: Forced — surgical method to achieve intraoperative hemostasis by a deep tissue electrocoagulation of 80 Watt voltage
  Arms: Forced

SUMMARY:
In a randomized clinical trial of 120 women undergoing large loop excision of the transformation zone (LLETZ)-conization for cervical dysplasia, two coagulation modes, spray versus forced coagulation, will be compared. The primary outcome of the study is time to complete hemostasis, secondary outcomes are intraoperative blood loss, postoperative pain, and postoperative bleeding complications.

DETAILED DESCRIPTION:
Intraoperative bleeding during large loop excision of the transformation zone (LLETZ)-conization can be achieved by two modes of electrocoagulation, spray coagulation and forced coagulation. Spray coagulation is a superficial coagulation mode, whereas forced coagulation is a deep tissue coagulation mode. It is unknown, whether spray or forced coagulation is superior regarding intraoperative hemostasis and other outcome Parameters such as postoperative bleeding and postoperative pain. Therefore, the investigator designed a randomized clinical trial of 120 women undergoing large loop excision of the transformation zone (LLETZ)-conization for cervical dysplasia, comparing the two coagulation modes, spray coagulation and forced coagulation, The primary outcome of the study is time to complete hemostasis measured in seconds, secondary outcomes are intraoperative blood loss measured as difference in serum hemoglobin pre- and postoperatively, postoperative pain according to a 10 step VAS scale, and postoperative bleeding complications, defined as necessity to intervene surgically for vaginal bleeding up to 14 days postoperatively. The study Population consists of women undergoing LLETZ-conization for histologically proven cervical dysplasia. The study hypothesis states that the difference in the mean time until complete hemostais will be at least 1/3 shorter in women randomized to spray coagulation. With a study Population of 120 women, this study has a power of >80% to detect a difference of 1/3 of the mean coagulation time until complete hemostais based on an anticipated mean time of 85 seconds.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven cervical dysplasia
* colposcopy Prior to LLETZ-conization
* informed consent
* no known hematologic disorder

Exclusion Criteria:

* significant language barrier
* a personal history of LLETZ-conization

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
time to complete intraoperative hemostasis | 120 seconds
  the time until complete hemostasis as judged by the surgeon has been achieved, will be measured in seconds

SECONDARY OUTCOMES:
postoperative pain | 5 hours
  patients will score their postoperative pain Level using a 10-step visual analogue scale (VAS) within 5 hours after surgery
postoperative complications | 14 days
  postoperative complications defined as the necessity to intervene surgically for vaginal bleeding within 14 days after surgery
intraoperative blood loss | 5 hours
  intraoperative blood loss will be measured using the difference in serum hemoglobin one day prior to surgery and within 5 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Ruhr University Bochum, Bochum, Germany

REFERENCES:
- [Result] Hilal Z, Mavrommati G, Foerster C, Rezniczek GA, Hefler LA, Tempfer CB. Spray Versus Forced Coagulation in Large Loop Excision of the Transformation Zone: A Randomized Trial. J Low Genit Tract Dis. 2016 Apr;20(2):169-73. doi: 10.1097/LGT.0000000000000177. PMID 26796660